CLINICAL TRIAL: NCT02666820
Title: Endoscopic Papillary Large Balloon Dilatation Versus Sphincterotomy +/- Mechanical Lithotripsy for Removal of Bile Duct Stones With a Mean Stone > 20 mm : A Randomized Controlled Study
Brief Title: Endoscopic Papillary Large Balloon Dilatation Versus Mechanical Lithotripsy for Large Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53-170-14-3-2
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Common Bile Duct Stones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Large balloon dilatation (Active Comparator): Patients underwent clearance of common bile duct stones using a papillary large balloon dilatation.
  Interventions: Procedure: Large balloon dilatation
- Mechanical lithotripsy (Active Comparator): Patients underwent clearance of common bile duct stones using a mechanical lithotripsy.
  Interventions: Procedure: Mechanical lithotripsy

INTERVENTIONS:
Procedure: Large balloon dilatation — After biliary sphincterotomy was performed with full extension to the full length of transverse fold. A 12, 15, 18 or 20 mm CRE-balloon was passed over guide wire and position across the papilla. The balloon was gradually inflated to the largest size of the bile duct stone and/or the bile duct diameter. When complete stone removal was unsuccessful , crossing over treatment was considered at the discretion of the endoscopists.
  Arms: Large balloon dilatation
Procedure: Mechanical lithotripsy — After biliary sphincterotomy was performed with full extension to the full length of transverse fold. A 3x6 cm Trapezoid Rx retrieval stone basket was used to capture the stone and crushing of stones was done when simple stone extraction failed to remove the stone. The stone fragments were then retrieved with a basket and/ or a retrieval balloon. When complete stone removal was unsuccessful , crossing over treatment was considered at the discretion of the endoscopists.
  Arms: Mechanical lithotripsy

SUMMARY:
Endoscopic sphincterotomy (EST) combined with large balloon dilation (LBD) has been increasingly accepted as alternative method for removal of large bile duct stones. However, there were limited studies comparing the efficacy of EST in combined with LBD to EST with mechanical lithotripsy (ML). The purpose of this study to compare the efficacy and safety of combined EST- LBD versus EST-ML in the removal of very large bile duct stones.

DETAILED DESCRIPTION:
The large common bile duct stones (CBDS) remains a therapeutic challenge in ERCPs. Large CBDS are generally refractory to be removed by EST and stone extraction balloons and or baskets. Traditional rescue therapy was the technique of stone fragmentation using ML. The previous reports have shown that EST with ML was successful in the fragmentation of large stones yielding stone clearance rate from 68 t0 79 %. EST-LBD has been shown favorable outcome in the treatment of large bile duct stone. A meta-analysis comparing the effectiveness and complications between EST-LBD and EST in the management of CBDS showed that EST-LBD was as effective as EST for the removal of large or difficult of CBDS in terms of stone clearance in the first ERCP session of 87.87 % vs. 84.15 % and overall clearance of 97.35 % vs. 96.35 % but EST-LBD was associated with fewer complications as well as reduced need for ML compared to EST. The efficacy of EST-ML versus EST-LBD as a therapy for relatively large CBDS, a mean stone size > 20 mm in currently not well defined. The investigators, herein, compared the efficacy and complications between EST followed by LBD or ML for the removal of CBDS > 15 mm with a mean stone size > 20 mm.

ELIGIBILITY:
Inclusion Criteria: -Patients with age>/= 18 years with confirmed or suspected CBDS at our institute were enrolled in the study.

* Informed consent was obtained in every patients prior to the procedure
* Patients were randomized to LBD or ML if they had CBD stone >/= 15 mm in shortest dimension or stone' size was disproportionate to the lower bile duct segment with a ratio of largest stone dimension/lower bile duct segment diameter > 50 % identified by a cholangiogram at ERCP.

Exclusion Criteria:-pregnant woman

* uncorrectable coagulopathy (INR >1.5 ), thrombocytopenia( platelet count < 50,000)
* concomitant intrahepatic duct stones
* ongoing acute pancreatitis or acute cholecystitis
* surgically altered anatomy (i.e. Billroth II or Roux-en-Y reconstruction)
* concomitant pancreatic or biliary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Complete stone clearance rate in the index ERCP | 24 hours
  The number of patients who was achieved complete stone clearance in the index ERCP

SECONDARY OUTCOMES:
Procedure time | 24 hours
  The procedure time was the time between insertion of the index device namely, a balloon or ML, and occlusion of cholangiogram
Complete stone clearance rate in the rescue therapy | 24 hours
  The number of patients who was achieved complete stone clearance in the rescue therapy
Complication rate | 30 days
  The number of patients who developed complications related procedure included pancreatitis, bleeding, perforation, cholangitis as defined and graded according to the consensus guideline and sedation related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Bancha Ovartlarnporn, MD., Study Director — NKC Institute of Gastroenterology and Hepatology, Faculty of Medicine, Prince of Songkla University, Hatyai, Songkhla, Thailand, 90110.
Locations (1):
- NKC Institue of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
The individual data of patients participating in the study are not available for public sharing since we did not obtain the consent to share the data of patient